CLINICAL TRIAL: NCT00245037
Title: A Phase I/II Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplant for the Treatment of Patients With Hematologic Malignancies Using Busulfan, Fludarabine and Total Body Irradiation
Brief Title: Busulfan, Fludarabine, and Total-Body Irradiation in Treating Patients Who Are Undergoing a Donor Stem Cell Transplant for Hematologic Cancer
Acronym: Bu Flu TBI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Maziarz, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000210; P30CA016058 (NIH); OHSU-HEM-05011-L (Other: OHSU Knight Cancer Institute); OHSU-210 (Other: OHSU IRB)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Precancerous Condition
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, breakpoint cluster region-Abelson (BCR-ABL) negative; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; chronic myelomonocytic leukemia; acute undifferentiated leukemia; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; stage I multiple myeloma; secondary acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precancerous Conditions; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Immunoglobulin Light-chain Amyloidosis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Monoclonal Gammopathy of Undetermined Significance; Congenital Abnormalities; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Busulfan; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Granulocyte Colony-Stimulating Factor; Phenytoin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI) (Experimental): Busulfan 3.2 mg/kg IV on day -5 Fludarabine 30 mg/m2/day x 3 (total dose 90 mg/m2, day -4 to day -2 TBI 200 centigray (cGy) x 1, day 0
  Interventions: Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: peripheral blood stem cell transplantation; Radiation: Total Body Irradiation (TBI); Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Phenytoin; Drug: Methotrexate

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — A population of lymphocytes therapeutically administered to a recipient individual who is genetically distinct from a donor of the same species.
Drug: busulfan — Busulfan is an alkylating chemotherapeutic agent which has been used in many high dose and reduced intensity regimens prior to allogeneic or autologous hematopoietic stem cell transplants. It is active in a wide variety of malignancies and in high-doses it is myeloablative.
  IV busulfan is available and diluted and administered per package insert guidelines.
Drug: cyclosporine — Cyclosporine is a cyclic polypeptide immunosuppressive agent. It blocks the calcium-dependent calcineurin-mediated nuclear localization of nuclear factor of activated T cells (NFAT) following T-cell activation, thereby inhibiting transactivation of key T-cell response genes including Interleukin 2 (IL-2) and Interleukin 4 (IL-4).
  - Starting on day -3, Cyclosporine (CSP) is given at a dose of 4.0 mg/kg p.o. b.i.d.
Drug: fludarabine phosphate — Fludarabine's active metabolite 2-fluoro-ara-A is an antimetabolite that inhibits DNA primase, DNA polymerase alpha and ribonucleotide nuclease.
  * Dosing: Days -4, -3 and -2: Fludarabine 30 mg/m2/day IV. Total dose equals 90 mg/m2.
  * Monitoring: Fludarabine level is not monitored.
  * Dose Adjustments: There are no provisions for fludarabine dose adjustments.
Drug: mycophenolate mofetil — Mycophenolate mofetil (MMF) is the morpholinyl ethyl ester of mycophenolic acid (MPA) and reversibly inhibits inosine monophosphate dehydrogenase, particularly the type II isoform that is more prominent in activated lymphocytes. As a result of the inhibition of de novo purine synthesis, proliferation of B- and T-lymphocytes is blocked and antibody production is inhibited.
  * Related Donors: MMF will be given daily at 15mg/kg q 12 hrs until day +28, then stop without tapering. Doses will be rounded to the nearest 250 mg (capsules are 250 mg).
  * Unrelated Donors: MMF will be given daily at 15mg/kg q 8 hrs until day +28, then given daily at 15mg/kg q 12 hours until day +56, then stop without tapering. Doses will be rounded to the nearest 250 mg (capsules are 250 mg).
Procedure: peripheral blood stem cell transplantation — Bone marrow transplantation (BMT) and peripheral blood stem cell transplantation (PBSCT) are procedures that restore stem cells that have been destroyed by high doses of chemotherapy and/or radiation therapy. There are three types of transplants:
  * In autologous transplants, patients receive their own stem cells.
  * In syngeneic transplants, patients receive stem cells from their identical twin.
  * In allogeneic transplants, patients receive stem cells from their brother, sister, or parent. A person who is not related to the patient (an unrelated donor) also may be used.
Radiation: Total Body Irradiation (TBI) — TBI is a form of radiotherapy used primarily as part of the preparative regimen for haematopoietic stem cell (or bone marrow) transplantation. As the name implies, TBI involves irradiation of the entire body, though in modern practice the lungs are often partially shielded to lower the risk of radiation-induced lung injury.
  * Toxicities: At the dosage used, side effects are not expected. Nevertheless, there may be fever, alopecia, parotitis, diarrhea, reversible skin pigmentation, mucositis and late effects including cataract formation, pulmonary damage, carcinogenesis, and sterilization.
  * Dosing: TBI will be given in one 200 cGy fraction from linear accelerator at a rate of 15-19 cGy/min.
Drug: Granulocyte colony-stimulating factor (G-CSF) — Granulocyte colony-stimulating factor (G-CSF or GCSF) is a colony-stimulating factor hormone. G-CSF is also known as colony-stimulating factor 3 (CSF 3).
  It is a glycoprotein, growth factor and cytokine produced by a number of different tissues to stimulate the bone marrow to produce granulocytes and stem cells. G-CSF then stimulates the bone marrow to release them into the blood.
  * Toxicities: At the dosage used, the most common side effect will be medullary bone pain.
  * Dosing: 5 mcg/kg/day given per institutional standards (on approximately days 10-15 or not at all).
Drug: Phenytoin — This drug is used to prevent seizures while on chemotherapy.
Drug: Methotrexate — Methotrexate is used to treat severe psoriasis (a skin disease in which red, scaly patches form on some areas of the body) that cannot be controlled by other treatments.

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and busulfan, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects of giving busulfan and fludarabine together with total-body irradiation and to see how well they work in treating patients who are undergoing a donor stem cell transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess safety and toxicity of the addition of busulfan added to an established fludarabine and low-dose total-body irradiation (TBI) conditioning regimen for non-myeloablative allogeneic transplantation in patients with hematologic malignancies. (Phase I)
* To assess the non-relapse mortality 1-year after conditioning with busulfan and fludarabine/TBI in patients with hematologic malignancies at moderate to high risk for graft rejection and/or relapse of underlying disease. (Phase II)

Secondary

* To assess overall survival 1-year survival. (Phase II)
* To assess the incidence of graft rejection. (Phase II)
* To assess the incidence of grade II-IV acute graft-vs-host disease (GVHD) and chronic extensive GVHD. (Phase II)
* To assess rates of disease progression and/or relapse-related mortality. (Phase II)
* To determine non-hematologic grade III-IV organ specific toxicity. (Phase II)

OUTLINE:

* Nonmyeloablative-conditioning regimen: Patients receive busulfan IV on day -5 and fludarabine IV over 30 minutes on days -4 to -2. Patients undergo total body irradiation on day 0.
* Allogeneic peripheral blood stem cell transplantation (PBSC): Patients undergo donor PBSC infusion on day 0.
* Graft-versus-host disease prophylaxis: Patients receive oral cyclosporine twice daily on days -3 to 56 followed by a taper to day 180. Patients with a related stem cell donor receive oral mycophenolate mofetil twice daily on days 0-28. Patients with an unrelated stem cell donor receive oral mycophenolate mofetil 3 times daily on days 0-28 followed by a taper twice daily to day 56. Patients with evidence of relapse or persistent disease may also receive up to 3 donor lymphocyte infusions.

PROJECTED ACCRUAL: A total of 225 patients will be accrued for this study; 25 patients accrued into the Phase I and 200 patients into Phase II.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematologic malignancy of 1 of the following high-risk types:

  * Acute lymphoblastic leukemia
  * Acute myeloid leukemia
  * Chronic myelogenous leukemia
  * Chronic lymphocytic leukemia
  * Myelodysplastic syndromes
  * Myeloproliferative disorder
  * Multiple myeloma
  * Plasma cell dyscrasias
  * Non-Hodgkin lymphoma
  * Hodgkin disease

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No liver failure
* No cirrhosis with evidence of portal hypertension
* No alcoholic hepatitis
* No esophageal varices
* No chronic hepatitis
* No other liver disease

Renal

* Not specified

Cardiovascular

* Left Ventricular Ejection Fraction (LVEF) > 35%
* No symptomatic coronary artery disease or cardiac failure requiring therapy

Pulmonary

* Diffusing capacity of lung for carbon monoxide (DLCO) > 30%
* Total lung capacity > 30%
* Forced expiratory volume in 1 second (FEV_1) > 30%
* No supplementary continuous oxygen

Other

* HIV negative
* No active nonhematologic malignancy except localized skin cancer
* No overt organ dysfunction

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2005-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Maziarz, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI): Busulfan 3.2 mg/kg IV on day -5 Fludarabine 30 mg/m2/day x 3 (total dose 90 mg/m2, day -4 to day -2 TBI 200 centigray (cGy) x 1, day 0
  Therapeutic allogeneic lymphocytes: A population of lymphocytes therapeutically administered to a recipient individual who is genetically distinct from a donor of the same species.
  Busulfan: Busulfan is an alkylating chemotherapeutic agent which has been used in many high dose and reduced intensity regimens prior to allogeneic or autologous hematopoietic stem cell transplants. It is active in a wide variety of malignancies and in high-doses it is myeloablative.
  IV Busulfan is available and diluted and administered per package insert guidelines.
  Cyclosporine: Cyclosporine is a cyclic polypeptide immunosuppressive agent. It blocks the calcium-dependent calcineurin-mediated nuclear localization of nuclear factor of activated T cells (NFAT) following T-cell activation, thereby inhibiting transactivation of key T-cell response genes including
Period: Overall Study
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Started | 147
Completed | 130 (17 participants died from infectious complications.)
Not Completed | 17
Not completed — Death | 17

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 81
  >=65 years | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 98
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS Scale:
  100 = Normal, no complaints, no evidence of disease. 90 = Able to carry on normal activity; minor signs or symptoms of disease. 80 = Normal activity with effort; some signs or symptoms of disease. 70 = Cares for self, unable to carry on normal activity or to do active work. 60 = Requires occasional assistance, but is able to care for most of his/her needs.
  50 = Requires considerable assistance and frequent medical care. 40-0 = Not eligible Population: Eight patients did not have KPS status available, which is why the values do not add up to the total number of participants.
  Participants
    number analyzed (Participants) | 139
    KPS ≥ 90 | 91
    KPS < 90 | 48
Pre-Transplant Disease Status [Count of Participants; unit: Participants]
  In Complete Remission | 85
  Not in Complete Remission | 62
Disease Risk Index (DRI) [Count of Participants; unit: Participants] — Population: DRI was unclassifiable in 3 patients.
  Participants
    number analyzed (Participants) | 144
    Low or intermediate | 93
    High or Very High | 51
HLA Match [Count of Participants; unit: Participants] — HLA Criteria:
  Related to the patient and genotypically or phenotypically HLA-identical (8/8). Single antigen mismatch (7/8) can be accepted if no other donor is available.
  OR
  Unrelated to the patient and HLA matched by molecular typing, allowing a single allele or antigen mismatch (7/8).
  Participants
    8/8 | 135
    7/8 | 12
Donor Relation [Count of Participants; unit: Participants]
  Related Sibling Donor | 39
  Unrelated Donor | 108
Cytomegalovirus (CMV) Status [Count of Participants; unit: Participants] — Population: Cytomegalovirus (CMV) status was unavailable in 7 patients.
  Participants
    number analyzed (Participants) | 140
    -/- recipient/donor | 22
    All other combinations | 118
Donor/Recipient Gender [Count of Participants; unit: Participants]
  F/F, M/M, M/F | 117
  F/M | 30

OUTCOME MEASURES:

1. Primary Outcome: Regimen-Related Toxicities
Description: Non-hematologic toxicities and adverse experiences ≥ Grade 3 occurrences measured up to day +100 using the NCI Common Toxicity Criteria for Adverse Events v3.0 (CTCAE). Infections and GVHD will be assessed up to 5 years post transplant. The following data represents the number of regimen-related, grade 3 and 4 toxicities that occurred in each category.
Time Frame: 5 years post-transplant
Measure: Number; unit: Toxicities
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
Toxicities
  Cardiac Disorders | 21
  Renal Disorders | 10
  Respiratory Disorders | 8
  CNS Disorders | 16
  Hepatic Disorders | 39
  General Disorders | 30

2. Primary Outcome: Non-relapse Mortality
Description: Percent of subjects with non-relapse mortality two years after conditioning with busulfan with fludarabine/200 cGy TBI in patients with hematologic malignancies at moderate to high risk for graft rejection and/or relapse of underlying disease.
Time Frame: Two years post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
Participants
  Year 1 | 27
  Year 2 | 33

3. Secondary Outcome: Overall Survival
Description: The percentage of overall patient survival (out of 147 participants) for Years 1, 2, 3 and 5.
Time Frame: Years 1, 2, 3 and 5
Measure: Number; unit: percentage of analyzed participants
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
percentage of analyzed participants
  Year 1 | 60
  Year 2 | 48
  Year 3 | 42
  Year 5 | 29

4. Secondary Outcome: Progression-Free Survival
Description: The percentage of progression-free patients (out of 147 participants) at Years 1, 2, 3, and 5.
  Definition of Disease Progression:
  MM/Plasma Cell: Increasing bone pain or increase in serum/urine monoclonal protein by 25%.
  CLL/NHL/HD: New sites of lymphadenopathy; ≥ 25% increase in lymph node size; Blood or bone marrow involvement with clonal B-cells; Increase of ≥ 25% bone marrow involvement; ≥ 25% increase in blood involvement with clonal B-cells.
  AML/ALL: Any incidence of relapse (>5% blasts) by evaluation of the bone marrow aspirate.
  CML: Inability to control platelet or granulocyte counts; Increase in baseline number of metaphases demonstrating the Ph+ chromosome by >25%; Any other new cytogenetic abnormality; Transformation to accelerated phase or blast crisis.
  MDS/MPD: Any evidence by morphologic or flow cytometric evaluation of the bone marrow aspirate of new blasts (>5%) or worsening cytopenia or cytogenetic evidence of recurrence.
Time Frame: Years 1, 2, 3, and 5
Measure: Number; unit: percentage of analyzed participants
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
percentage of analyzed participants
  Year 1 | 48
  Year 2 | 39
  Year 3 | 35
  Year 5 | 29

5. Secondary Outcome: Relapse Mortality
Description: The percentage of patients (out of 147 participants) who relapsed at Years 1 and 2. Relapse is defined as the presence of >5% blasts by morphology on a post-transplant bone marrow aspirate.
Time Frame: Years 1 and 2
Measure: Number; unit: percentage of analyzed participants
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
percentage of analyzed participants
  Year 1 | 13
  Year 2 | 20

6. Secondary Outcome: Acute Graft-Versus-Host Disease (aGVHD) Outcome
Description: Grading of Acute GVHD:
  Severity of Individual Organ Involvement:
  Skin
  * 1 a maculopapular eruption involving less than 25% of the body surface
  * 2 a maculopapular eruption involving 25-50% of the body surface
  * 3 generalized erythroderma
  * 4 generalized erythroderma with bullous formation and/or with desquamation Liver
  * 1 bilirubin 2.0-3.0mg/100mL
  * 2 bilirubin 3-5.9mg/100mL
  * 3 bilirubin 6-14.9mg/100mL
  * 4 bilirubin >15mg/100mL Gut Diarrhea is graded +1 to +4 in severity. Nausea/vomiting and/or anorexia caused by GVHD is assigned as +1 in severity Diarrhea
  * 1 <1000mL of liquid stool/day
  * 2 >1,000mL of stool/day
  * 3 >1,500mL of stool/day
  * 4 2,000mL of stool/day, severe abdominal pain, with or without ileus
  Severity of GVHD:
  Grade 1 +1 to +2 skin rash; No gut or liver involvement Grade 2 +1 to +3 skin rash;+1 GI involvement and/or +1 liver
Time Frame: Day 100, Month 6
Population: This is cumulative incidence of grades 2-4 aGVHD at 100 days and at 6 months. Out of the total number of participants, grades 2-4 aGVHD occurred in 79 patients.
Measure: Number; unit: percentage of analyzed participants
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
percentage of analyzed participants
  Day 100 | 55
  Month 6 | 60

7. Secondary Outcome: Chronic Graft-Versus-Host Disease (cGVHD) Outcome
Description: Grading of Chronic GVHD:
  Limited: Localized skin involvement and/or hepatic dysfunction due to chronic GVHD
  Extensive:
  One or more of the following:
  Generalized skin involvement Liver histology showing chronic aggressive hepatitis, bridging necrosis or cirrhosis Involvement of the eye: Schirmer's test with <5 mm wetting Involvement of minor salivary glands or oral mucosa demonstrated on labial biopsy Involvement of any other target organ
  Chronic GVHD Severity:
  Mild: Signs and symptoms of cGVHD do not interfere substantially with function and do not progress once appropriately treated with local therapy or standard systemic therapy.
  Moderate: Signs and symptoms of cGVHD interfere somewhat with function despite appropriate therapy or are progressive through first line systemic therapy.
  Severe: Signs and symptoms of cGVHD limit function substantially despite appropriate therapy or are progressive through second line systemic therapy
Time Frame: Years 1, 2 and 3
Population: This is a cumulative incidence of cGVHD at 1 year, 2 years, and 3 years. A total of 99 patients (out of 147) developed cGVHD, 86 patients (87%) with extensive stage cGVHD and 13 patients (13%) with limited stage cGVHD.
Measure: Number; unit: percentage of analyzed participants
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Number analyzed (Participants) | 147
percentage of analyzed participants
  Year 1 | 64.6
  Year 2 | 66
  Year 3 | 67.3

ADVERSE EVENTS:
Time Frame: Non-hematologic toxicities and adverse experiences ≥ Grade 3 will be assessed up to day +100 using the NCI Common Toxicity Criteria for Adverse Events v3.0 (CTCAE). Infections and GVHD will be assessed up to 5 years post transplant.
Arm/Group | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI)
Serious Adverse Events (participants affected / at risk) | 59/147
Other Adverse Events (participants affected / at risk) | 52/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI) (N=147)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 — Related to regimen
Pericardial effusion (Cardiac disorders) | 2 — Related to regimen
Atrial fibrillation/flutter (Cardiac disorders) | 3 — Related to regimen
Left ventricular dysfunction (Cardiac disorders) | 1 — Related to regimen
Respiratory pulseless electrical activity (PEA) arrest (Cardiac disorders) | 1 — Related to regimen
Event associated with CsA (Renal and urinary disorders) | 1 — Related to regimen
Cryptogenic organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — Related to regimen
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — Related to regimen
CsA toxicity (Nervous system disorders) | 5 — Related to regimen
Posterior-reversible encephalopathy syndrome (Nervous system disorders) | 2 — Related to regimen
Veno-occlusive disease (Hepatobiliary disorders) | 1 — Related to regimen
Iron overload (General disorders) | 1 — Related to regimen
Steroid myopathy (General disorders) | 3 — Related to regimen
Hemolysis (General disorders) | 5 — Related to regimen
ABO incompatability (General disorders) | 1 — Related to regimen
Bleeding (General disorders) | 2 — Related to regimen
Thrombosis/deep vein thrombosis (General disorders) | 5 — Related to regimen
Thrombotic thrombocytopenic purpura (TTP) (General disorders) | 1 — Related to regimen
Refractory ascites (General disorders) | 1 — Related to regimen
Ogilvie's syndrome (General disorders) | 1 — Related to regimen
Fractures/musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 — Related to regimen
Death Caused by Bacterial Infection (Infections and infestations) | 7 — Unrelated to regimen
Death Caused by Fungal Infection (Infections and infestations) | 3 — Unrelated to regimen
Death Caused by Sepsis/Septic Shock (Infections and infestations) | 3 — Unrelated to regimen
Death Caused by Viral Infection (Infections and infestations) | 3 — Unrelated to regimen
Death Caused by Nonspecified Pneumonia (Infections and infestations) | 1 — Unrelated to regimen
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan (Bu), Fludarabine (Flu), Total Body Iradiation (TBI) (N=147)
Neutropenic fever (Infections and infestations) | 14 — Unrelated to Regimen
Hyperbilirubinemia or transaminitis (Hepatobiliary disorders) | 38 — Related to regimen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes